CLINICAL TRIAL: NCT04396002
Title: Glaucoma, Visual Field Loss, and Their Association With Life Space in Older Adults
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lyne Racette, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 300001552; 5P30AG022838-14 (NIH)
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Dark Adaptation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Open-Angle Glaucoma: Patients diagnosed with primary open-angle glaucoma.
  Interventions: Diagnostic Test: Life Space Questionnaire; Diagnostic Test: Low Luminance Questionnaire; Diagnostic Test: Contrast sensitivity under dim illumination; Diagnostic Test: Visual field under dim illumination (MAIA); Diagnostic Test: Macular Pigment Optical Density (MPOD); Diagnostic Test: Dark Adaptation
- Control: Participants with healthy eyes.
  Interventions: Diagnostic Test: Life Space Questionnaire; Diagnostic Test: Low Luminance Questionnaire; Diagnostic Test: Contrast sensitivity under dim illumination; Diagnostic Test: Visual field under dim illumination (MAIA); Diagnostic Test: Macular Pigment Optical Density (MPOD); Diagnostic Test: Dark Adaptation

INTERVENTIONS:
Diagnostic Test: Life Space Questionnaire — This 9-item questionnaire is interested in finding out how much a person gets out and about and the spatial extent of the person's typical life space, i.e., what is the usual range of places in which the person engages in activities within the designated time frame.
Diagnostic Test: Low Luminance Questionnaire — This 32-item questionnaire is interested in finding out problems that involve vision under different lighting conditions or feelings that people have about your vision under different lighting conditions.
Diagnostic Test: Contrast sensitivity under dim illumination — Participants will be presented with visual targets of different contrast under dim illumination and asked to report when they see the target.
Diagnostic Test: Visual field under dim illumination (MAIA) — Sensitivity in the central visual area will be assessed under dim illumination
Diagnostic Test: Macular Pigment Optical Density (MPOD) — Participants will be asked to look at a fixation target and the density of their macular pigment will be assessed.
Diagnostic Test: Dark Adaptation — After adapting to a dark environment, participants will be exposed a bright flask of light. the time needed for them to recover their sensitivity will be measured.

SUMMARY:
Mobility refers to a person's purposeful movement through the environment from one place to another and can be conceptualized as a continuum from bed bound (immobility) on one extreme to making excursions to distant locations on the other extreme. Primary open-angle glaucoma (POAG) is a chronic, progressive optic neuropathy that can lead to gradual loss of vision in the peripheral field and central vision. Older adults with POAG have an increased risk for motor vehicle collisions and falls. Moreover, existing studies suggest that patients with POAG exhibit more postural sway while standing as measured by a balance platform and also tend to walk more slowly than those who are normally sighted and free of ocular disease. While these disturbances likely influence mobility, there has been little research directly assessing the impact of POAG on mobility. This study will assess the impact of POAG on life space (one aspect of mobility) and will determine whether difficulties with life space are associated with difficulties experienced under conditions of dim lighting.

DETAILED DESCRIPTION:
Aim 1: To determine whether differences exist between people with healthy eyes and patients with POAG in seeing under dim illumination (Low Luminance Questionnaire) and to determine whether such differences are associated with life space.

Aim 2: To determine whether differences exist between people with healthy eyes and patients with POAG in seeing under dim illumination (objective measures of visual function) and to determine whether such differences are associated with life space.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Participants that are enrolled in the Early Detection of Glaucoma Progression using a Novel Individualized Approach (IRB-300000301) or in the African Descent and Glaucoma Evaluation (ADAGES) IV: Alterations of the Lamina Cribrosa in Progression (IRB-161115004).

Exclusion Criteria (Patients):

* Not being enrolled in one of the following two NIH-funded studies: 1. African Descent and Glaucoma Evaluation (ADAGES) IV: Alterations of the lamina cribrosa in progression (EY026574) or 2. Early detection of glaucoma progression using a novel individualized approach (EY025756)

Inclusion Criteria (Controls):

* No diagnosis of eye disease

Exclusion Criteria (Controls):

* Cognitive impairment that would preclude ability to take the tests

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients:
  Participants that are enrolled in the Early Detection of Glaucoma Progression using a Novel Individualized Approach (IRB-300000301) or in the African Descent and Glaucoma Evaluation (ADAGES) IV: Alterations of the Lamina Cribrosa in Progression (IRB-161115004).
  Controls:
  Participants with healthy eyes will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of life space measured with the Life Space Questionnaire | Through study completion, an average of 1 year
  The Life Space Questionnaire is a 9-item questionnaire that assesses how much a person gets out and about and the spatial extent of the person's typical life space, i.e., what is the usual range of places in which the person engages in activities within the designated time frame. Patients are asked to respond either Yes or No.
Assessment of vision under low luminance conditions | Through study completion, an average of 1 year
  The Low Luminance Questionnaire is a 32-item questionnaire that assesses how participants see under dim illumination and how well they can perform different tasks (e.g. reading, driving). Patients are asked to select a response among different choices on a Likert scale that ranges from 1 to 5, 1 to 6, 1 to 7, or 1 to 8 depending on the question. A response of "1" indicates that the participant experiences no difficulty while increasingly higher numbers indicate increasing amounts of difficulty.
Differences in contrast sensitivity functions between controls and patients | Through study completion, an average of 1 year
  Participants will be presented with targets of different spatial frequency at different contrasts. Their sensitivity at each spatial frequency will be recorded/
Differences in dark adaptation between controls and patients | Through study completion, an average of 1 year
  Once participants have adapted to a dark environment, they will be exposed to a bright flash of light. The time needed to recover their visual sensitivity will be measured (rod-intercept time).
Differences in visual sensitivity under dim illumination between controls and patients | Through study completion, an average of 1 year
  Participants will be presented with targets at different locations in their visual fields under dim illumination.
Differences in Macular Pigment Optical Density between controls and patients | Through study completion, an average of 1 year
  Participants will fixate on a target while their MPOD is assessed. The MPOD is measured using the Heidelberg optical coherence tomography (OCT) MPOD module. Two different light sources are directed to the back of the eye. The light is reflected back and the OCT/MPOD computes the difference in the reflectance of the two lights which is an estimate of the density of macular pigment.
Assessment of the relationship between each the measure of visual function and life space | Through study completion, an average of 1 year
  The relationship between each of the measures of visual function (dark adaptation, contrast sensitivity functions, visual fields under dim illumination, and MPOD) and life space (Life Space Questionnaire will be assessed.
Assessment of the relationship between each the measure of visual function and self-reported visual function under dim illumination | Through study completion, an average of 1 year
  The relationship between each of the measures of visual function (dark adaptation, contrast sensitivity functions, visual fields under dim illumination, and MPOD) and self-reported visual performance under dim illumination (Low Luminance Questionnaire) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Lyne Racette, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No